CLINICAL TRIAL: NCT06747143
Title: "Study of Immunological Biomarkers in Response to Probiotic Intake"
Brief Title: Short-term Immunomodulatory Effects of Lactobacillus Casei DN-114001: Impacts on Gut Microbiota Composition and Systemic Immune Biomarkers in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valladolid (Other)
Collaborators: Danone Global Research & Innovation Center (Industry)
Responsible Party: Principal Investigator, Alfredo Corell, Prof. Dr., University of Valladolid
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PROBIOINMUNE2003
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Immune Modulation
Keywords: lactobacillus casei

STUDY DESIGN:
Intervention Model Description: Sequential intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Healthy subjects
  Interventions: Dietary Supplement: Lactobacillus casei DN-114001

INTERVENTIONS:
Dietary Supplement: Lactobacillus casei DN-114001 — Probiotic
  Other Names: Actimel

SUMMARY:
The study included 21 adult participants, aged 19-46 years (19 female participants and 2 male participants). The selection criteria included the following parameters: Body Mass Index (BMI), calculated as weight (kg) divided by height squared (m²), between 18.5 and 29.99; Waist-to-Hip Ratio with thresholds set at >0.90 for males and >0.85 for females for individuals with normal weight (eutrophic); percentage of body fat: Considered within normal range if <30% for individuals with normal weight. Standard biochemical and anthropometric measurements were carried out to all the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 18.5 and 29.99;
* Waist-to-Hip Ratio with thresholds set at >0.90 for males and >0.85 for females for individuals with normal weight (eutrophic)
* Percentage of body fat: Considered within normal range if <30% for individuals with normal weight.

Ages: 19 Years to 46 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2013-02-01; Primary Completion 2013-04 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Fecal flora cultures (Count of colonies/mL) | From enrollment to the end of treatment at 45 days weeks, every 15 days
  Relative amount of colonies (CFU) of Escherichia coli, Clostridium species and Lactobacillus
Serum immunoglobulins | From enrollment to the end of treatment at 45 days weeks, every 15 days
  Serum concentration of G, A, M, and G subclasses, as well as the complement C3 and C4 factors,
Lymphocyte Subpopulations | From enrollment to the end of treatment at 45 days weeks, every 15 days
  Concentration of T Lymphocytes: CD3, CD4, CD8, CD45 RA, and CD45 RO (distinguishing between helper T cells, cytotoxic T cells, and naïve or memory subsets within each group). ii) B Lymphocytes: CD19; iii) NK Cells: CD16 and CD56.

IPD SHARING:
Plan to Share IPD: No
Not needed